CLINICAL TRIAL: NCT06511232
Title: Intraosseous Morphine Administration During Anterior Cruciate Ligament Reconstruction: a Randomized Control Trial
Brief Title: Intraosseous Morphine Administration During Anterior Cruciate Ligament Reconstruction
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: The Methodist Hospital Research Institute (Other)
Responsible Party: Principal Investigator, Robert A. Jack, Assistant Professor of Clinical Orthopedic Surgery, Academic Institute, The Methodist Hospital Research Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: PRO00037918
Record Dates: First submitted 2024-07-02; First posted 2024-07-19 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-08

CONDITIONS: Anterior Cruciate Ligament Tear; Anterior Cruciate Ligament Injuries; Anterior Cruciate Ligament Rupture
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries | interventions — Morphine

STUDY DESIGN:
Intervention Model Description: This study is a single-blind randomized controlled trial with two arms, 1) Intervention and 2) control. The intervention group will receive an intraosseous (IO) injection of 10mg of morphine mixed with up to 100mg of saline into the tibial tubercle. The control group will receive the standard of care treatment, which is no IO injection. The subjects' post-operative pain levels, pain medication consumption, side effects to pain medications, and range of motion will be recorded for 14 days following surgery. Additionally, patient reported outcomes will be tracked via surveys prior to surgery and 2, 6, and 12-weeks following surgery.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intraosseous Injection of Morphine (Experimental): The intervention group will receive an intraosseous (IO) injection of 10mg of morphine mixed with up to 100mg of saline into the tibial tubercle during a standard ACL reconstruction.
  Interventions: Drug: Intraosseous Morphine
- Standard of Care Morphine Administration (No Intervention): The control group will receive the standard of care treatment, which is no IO injection during a standard ACL reconstruction.

INTERVENTIONS:
Drug: Intraosseous Morphine — More recently, intraosseous infusion of analgesics and antibiotics has gained traction in the total joint arthroplasty literature. In knee arthroplasty patients, the combination of a spine and adductor canal block with an intraosseous infusion of morphine into the tibial tubercle prior to incision yielded lower pain in the immediate postoperative period and at 2 weeks, less pain medication use, and significantly better patient-reported outcomes while also reducing systemic opioid exposure in the early postoperative period compared to the spine and adductor block alone.3 No study to date in the available literature has evaluated the efficacy of intraosseous morphine infusion in managing acute postoperative pain in patients undergoing ACL reconstruction with bone-patellar tendon-bone autograft, so that is the intended evaluation point with this project.
  Other Names: Duramorph; Astramorph PF; Infumorph
  Arms: Intraosseous Injection of Morphine

SUMMARY:
The purpose of this study is to determine if intraosseous (IO) morphine decreases pain and post-operative opioid use in patients undergoing anterior cruciate ligament (ACL) reconstruction.

ELIGIBILITY:
Inclusion Criteria:

* Patients of the IRB approved surgeon(s) undergoing ACL reconstruction with bone-to-bone (BTB) autograft
* Patients aged between 18-40 years old at the time of surgery

Exclusion Criteria:

* Patients undergoing ACL reconstruction with any other type of autograft or allograft other than BTB
* Patients younger than 18 years old or older than 40 years old
* Patients undergoing meniscal root repair or any other repair that changes their weight-bearing status
* Patients with a history of substance abuse
* Vulnerable populations
* Patients on chronic pain medication within the last 6 months
* BMI >/= 35
* Allergy to morphine
* Unwilling to participate
* Any additional reason the PI deems reasonable

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 84 (Estimated)
Dates: Start 2024-08-19 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2029-07-31 (Estimated)

PRIMARY OUTCOMES:
Patient Pain Levels in the Post-Operative Period as assessed by a patient-reported post operative symptom journal. | 2 weeks postop, 6 weeks postop, 12 weeks postop
  The study will measure patient-reported levels of pain on a daily basis (for a total of two weeks) with a symptom journal, which will ask patients to report on a variety of pain-related outcomes including levels of pain throughout different times of day, levels of nausea throughout different times of the day, and what pain medication(s) they are taking and at what time.
Changes in Post-Operative Opioid Use | 2 weeks postop
  To examine if the use of IO morphine will result in different levels of post-operative opioid use compared to SOC administration of morphine. This outcome will be assessed utilizing the daily symptom journal which will ask patients to complete daily logs of the pain medication that they take (what kind, what dose, when they took it, etc.) for two weeks following their operation.
Patient Pain Levels in the Post-Operative Period as assessed by the Lysholm Knee Survey | 2 weeks postop, 6 weeks postop, 12 weeks postop
  Participants will be asked to complete the Lysholm Knee survey at 2, 6, and 12 weeks postop which will assess patient progress following surgery such as pain, swelling, climbing stairs, using a crutch, etc. The Lysholm scale consists of eight items with each question response being assigned an arbitrary score on an increasing scale. The total score is the sum of each response to the eight questions and may range from 0-100 where higher scores indicate a better outcome with fewer symptoms or disability.

SECONDARY OUTCOMES:
Patient Range of Motion in the Post-Operative Period as assessed by the KOOS, JR Knee Survey | Preop, 2 weeks postop, 6 weeks postop, 12 weeks postop
  Patients will complete the KOOS, JR. Knee Survey to self-report their level of difficulty/pain (from none to extreme) certain movements have caused them. KOOS, JR is scored by summing the raw response (range 0-28) and then converting it to an interval score. The interval score ranges from 0 to 100 where 0 represents total knee disability and 100 represents perfect knee health.
Patient Activity Level in the Post-Operative Period as assessed by the Tegner scale. | Preop, 2 weeks postop, 6 weeks postop, 12 weeks postop
  Patients will complete the Tegner Activity Level Survey which will ask them to self-report their pre-operative and post-operative level of activity. The rating system scores a person's activity level between 0 and 10, where 0 is "sick leave or disability pension because of knee problems" and 10 is "participation in competitive sports such as soccer at a national or international elite level." As such, a higher score reflects better outcomes on this measure.
Patient Range of Motion in the Post-Operative Period as assessed by the Lysholm Knee Survey | 2 weeks postop, 6 weeks postop, 12 weeks postop
  The Lysholm Knee Survey will ask specific questions with a variety of responses to reflect movement-ability responses such as the use of a cane, the presence of a limp, squatting, climbing stairs, etc.The Lysholm scale consists of eight items with each question response being assigned an arbitrary score on an increasing scale. The total score is the sum of each response to the eight questions and may range from 0-100 where higher scores indicate a better outcome with fewer symptoms or disability.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Jack, MD, Principal Investigator — The Methodist Hospital Research Institute
Locations (1):
- Houston Methodist Research Institute, Houston, Texas, United States